CLINICAL TRIAL: NCT04533594
Title: Improving Self-efficacy Through A Telenovela Intervention for Caregivers of Patients Receiving Hospice Care: Feasibility Study
Brief Title: Improving Self-Efficacy Through a Telenovela: Feasibility Study
Acronym: NOVELA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Colorado, Denver (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00256812; U2CNR014637 (NIH)
Record Dates: First submitted 2020-08-28; First posted 2020-08-31 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: videos; hospice family caregivers; education; telenovelas; self-efficacy; anxiety; feasibility
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single group pretest-posttest design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NOVELA (Experimental): Hospice family caregivers will work with the interventionist to use a web-enabled device (computer, smartphone or tablet) to access and view the video (3-6 mins) over the course of 4 hospice telehealth visits.
  Interventions: Behavioral: NOVELA

INTERVENTIONS:
Behavioral: NOVELA — The family caregivers that consent to participate will work with the interventionist to use a web-enabled device (computer, smartphone or tablet) to access and view the telenovela video (one of four episodes, each 3-6 mins) over the course of 4 hospice visits (one episode per visit). All four visits will be in person using telehealth via video-conferencing. The number of visits is based on the number of videos which content is prioritized based on previous work. The interventionist will introduce the purpose and topic of the video, facilitate video viewing and then elicit clarifying questions and reinforce main message.

SUMMARY:
In the NOVELA intervention, hospice care will be enhanced with the telenovela videos for hospice family caregivers (HFCG) education during weekly hospice visits to prepare caregivers for proper use of hospice support and healthcare services

DETAILED DESCRIPTION:
Telenovela is a television drama or soap opera that can be used to lead viewers to contemplate and discuss critical issues through video storytelling. Prior work showed informational telenovelas had a positive effect on Latino family caregivers' attitudes toward end-of-life (EOL) care services. The role of videos in hospice and palliative care shows significant promise, underscoring the videos as a mode of education for family caregivers that could potentially enhance caregiver's self-efficacy, decrease caregiver's anxiety, and reduce burnout. Despite the value of video education, many programs have failed to provide engaging material.

Based on input from HFCG, the investigators have produced a bilingual (Spanish and English version) four chapter telenovela video series (To Care/ El privilegio de cuidar) as part of NCI funded diversity supplement study. Founded upon extensive preliminary work, To Care portrays the journey of one hospice family as the family struggle with the hospice decision, pain management, decision-making, and finally the dying process. Averaging only 4:65 minutes, each chapter addresses one of these problems, validating family experiences and identifying potential solutions. Based on this work and interviews with hospice staff the investigators have built an intervention, NOVELA, to disseminate telenovelas to family caregivers in hospice agencies. The investigators will test the feasibility of NOVELA delivery in the hospice setting and evaluate efficacy of the intervention. The overall expectation is that NOVELA will improve self-efficacy thus lowering anxiety in hospice family caregivers. This proposal has the following aims:

* Specific Aim 1: To pilot test the feasibility and acceptability of integrating NOVELA with hospice care for family caregivers of hospice patients
* Specific Aim 2: To investigate the preliminary efficacy of integrating NOVELA with hospice care for family caregivers of hospice patients

ELIGIBILITY:
Inclusion Criteria:

* Identified family caregiver of patients enrolled in hospice
* Caregivers must be over the age of 18
* Without cognitive impairment
* With access to wireless device and internet.

Exclusion Criteria:

* HFCG of patients that are actively dying
* Caregivers younger than 18 years
* With cognitive impairment
* Without internet access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DULCE CRUZ-OLIVER, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Univeristy, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data will be submitted to the Palliative Care Research Cooperative (PCRC) data repository at the end of pilot study.
Supporting Information: CSR
Time Frame: One year after completion or after publication of results and data will be available for an unknown duration of time.
Access Criteria: Investigators may request access to the de-identified PCRC Data Repositories for secondary data analysis. Each request must be submitted in writing, must identify the research question that will be addressed, and must specify the data elements that are requested. Each request must also include a data security plan and explanation of how and for how long the data will be stored and who will have access to the data. The PCRC, and when applicable the Study Principal Investigator (PI), reviews all data requests. If all requirements are adequately met, arrangements are made to transfer the data in the most efficient, secure,and affordable manner to the requesting investigator.
URL: http://palliativecareresearch.org/

REFERENCES:
- [Background] Crist JD, Pasvogel A, Hepworth JT, Koerner KM. The impact of a telenovela intervention on use of home health care services and Mexican American older adult and caregiver outcomes. Res Gerontol Nurs. 2015 Mar-Apr;8(2):62-76. doi: 10.3928/19404921-20150105-02. Epub 2015 Jan 16. PMID 25594360
- [Background] Cruz-Oliver DM, Malmstrom TK, Fernandez N, Parikh M, Garcia J, Sanchez-Reilly S. Education Intervention "Caregivers Like Me" for Latino Family Caregivers Improved Attitudes Toward Professional Assistance at End-of-life Care. Am J Hosp Palliat Care. 2016 Jul;33(6):527-36. doi: 10.1177/1049909115584315. Epub 2015 May 27. PMID 26019262
- [Background] Washington KT, Oliver DP, Benson JJ, Rolbiecki AJ, Jorgensen LA, Cruz-Oliver DM, Demiris G. Factors influencing engagement in an online support group for family caregivers of individuals with advanced cancer. J Psychosoc Oncol. 2020 May-Jun;38(3):235-250. doi: 10.1080/07347332.2019.1680592. Epub 2019 Nov 6. PMID 31690247
- [Background] Cruz-Oliver DM, Abshire M, Budhathoki C, Oliver DP, Volandes A, Smith TJ. Reflections of Hospice Staff Members About Educating Hospice Family Caregivers Through Telenovela. Am J Hosp Palliat Care. 2021 Feb;38(2):161-168. doi: 10.1177/1049909120936169. Epub 2020 Jul 8. PMID 32638608
- [Derived] Cruz-Oliver DM, Blinka MD, Milner GE, Nelson KE, Bugayong M, Durkin N, Gallo JJ, Oliver DP, Abshire Saylor M. A Mixed-Methods Analysis of Response to NOVELA Among Hospice Family Caregivers. Am J Hosp Palliat Care. 2025 Sep 12:10499091251371149. doi: 10.1177/10499091251371149. Online ahead of print. PMID 40938148
- [Derived] Cruz-Oliver DM, Abshire Saylor M, Nelson KE, Milner GE, Blinka MD, Durkin N, Budhathoki C, Parker-Oliver D, Smith TJ. Hospice Family Caregiver Perceptions of Benefits and Challenges of a Telenovela Educational Intervention. J Palliat Med. 2022 Jun;25(6):945-951. doi: 10.1089/jpm.2021.0628. Epub 2022 Apr 20. PMID 35446674

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 participants had their "loved one" died before starting intervention
Period: Overall Study
Arm/Group | NOVELA
Started | 59 (Participants who completed baseline survey)
Started Intervention (N=6 participants had their loved one died before being able to start intervention) | 53 (Participants who started intervention after completion of baseline survey)
Completed Final Survey | 44 (Participants who completed second survey up to 8 weeks after baseline.)
Completed (N=20 participants had their loved one died before being able to complete the intervention.) | 33 (Participants that observed all 4 videos and, therefore, completed intervention)
Not Completed | 26
Not completed — Death | 26

BASELINE CHARACTERISTICS:
Arm/Group | NOVELA
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 40
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 59
Education [Count of Participants; unit: Participants] — Self-reported highest education
  Participants
    Primary or secondary school | 16
    College, equivalent and advanced | 42
    Did not report | 1
Marital Status [Count of Participants; unit: Participants] — Self-reported marital status
  Participants
    Married and/or have a partner | 44
    Divorced and/or separated | 9
    Widowed | 1
    Other (never married or unknown | 5
Relationship to patient [Count of Participants; unit: Participants] — Self-reported participant relationship to hospice patient
  Participants
    Child | 29
    Parent | 4
    Spouse or Life Partner | 15
    Other(grandchild, grandparent, friend, sibling, son/daughter-in-law and nephew). | 11
Hospice diagnosis [Count of Participants; unit: Participants] — Caregiver-reported diagnosis for hospice admission
  Participants
    Cancer | 19
    Cardiovascular | 11
    Neurologic | 14
    Other (multi-system, infectious and renal. ) | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in HFCG Anxiety Before and After NOVELA as Assessed by the Generalized Anxiety Disorder 7-item Scale
Description: Generalized Anxiety Disorder 7-item (GAD-7) scale. Family caregiver indicate the frequency they have been bothered by generalized anxiety. 7-items, scale 0-3, score range 0-21; higher scores reflect higher anxiety.
  Final score was collected up to 8 weeks from baseline.
Time Frame: Baseline and up to 8 weeks
Population: Only 43 participants had baseline and up to 8 weeks data. The goal was to analyze data for participants who had scores for the baseline and final assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NOVELA
Number analyzed (Participants) | 43
score on a scale
  Baseline | 8.63 (5.41)
  Final | 7.67 (4.77)

2. Primary Outcome: Change in HFCG Self-efficacy Before and After NOVELA as Assessed by the Caregiver Self-Efficacy Scale
Description: Caregiver Self-Efficacy Scale (CaSES) - 21-items, scale 1-4, score range 1-4; higher scores reflect higher self-efficacy.
  Final score was collected up to 8 weeks from baseline.
Time Frame: Baseline and up to 8 weeks
Population: We had 44 participants that completed baseline and up to 8 weeks. The goal was to analyze data for participants who had scores for the baseline and final assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NOVELA
Number analyzed (Participants) | 44
score on a scale
  Baseline | 3.01 (0.47)
  Final score | 3.05 (0.40)

3. Secondary Outcome: Change in HFCG Satisfaction During and After NOVELA as Assessed by a Single-item Satisfaction Question
Description: Single-item satisfaction question related to HFCG satisfaction with intervention. Investigator developed Likert scale item scored from 1 to 5 where 1 = "Not satisfied" and 5 = "Very satisfied".
  First score was at 2 weeks and final score was up to 6 weeks from first score assessment.
Time Frame: 2 weeks and up to 6 weeks
Population: We had first and final score of 35 participants. The goal was to analyze data for participants who had scores for the first and final assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NOVELA
Number analyzed (Participants) | 35
score on a scale
  First score | 4.02 (1.06)
  Final score | 4.26 (0.89)

ADVERSE EVENTS:
Description: Adverse events data was not collected.
Arm/Group | NOVELA
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT04533594/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT04533594/SAP_001.pdf